CLINICAL TRIAL: NCT01600807
Title: Phase I/II Trial of OSI-906 in Combination With Gemcitabine and Erlotinib in Patients With Metastatic Ductal Adenocarcinoma of the Pancreas
Brief Title: OSI-906 With Gemcitabine and Erlotinib for Metastatic Ductal Adenocarcinoma of the Pancreas
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was pending major changes and was on hold, pending activation; administratively withdrawn; will be submitted as a new protocol if study is revised.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Brian Wolpin, MD, MPH, Overall PI, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-148
Record Dates: First submitted 2011-08-08; First posted 2012-05-17 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Pancreatic Cancer, Metastatic
Keywords: Metastatic; Pancreas; Cancer; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms; Adenocarcinoma | interventions — Gemcitabine; Erlotinib Hydrochloride; 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine, Erlotinib, OSI-906 (Experimental): Experimental treatment arm
  Interventions: Drug: Gemcitabine, Erlotinib, OSI-906
- Gemcitabine, Erlotinib (Active Comparator): Standard treatment arm
  Interventions: Drug: Gemcitabine, Erlotinib

INTERVENTIONS:
Drug: Gemcitabine, Erlotinib, OSI-906 — Gemcitabine 1000 mg/m2 d1,8,15; Erlotinib 100 mg QD, OSI-906 dose to be determined BID
  Other Names: Gemzaar; Tarceva
  Arms: Gemcitabine, Erlotinib, OSI-906
Drug: Gemcitabine, Erlotinib — Gemcitabine 1000 mg/m2 d1,8,15; Erlotinib 100 mg QD
  Other Names: Gemzaar; Tarceva
  Arms: Gemcitabine, Erlotinib

SUMMARY:
OSI-906 is a new drug that may stop cancer cells from growing abnormally. This drug has been used in other research studies and information from those suggests that OSI-906 may help block cell receptors involved in tumor growth.

Gemcitabine and erlotinib are used as standard treatment for pancreatic cancer. In this research study, the investigators are looking for the highest dose of OSI-906 that can be given safely in combination with gemcitabine and erlotinib. This dose will then be given together with gemcitabine and erlotinib to a further group of patients with pancreatic cancer.

DETAILED DESCRIPTION:
This study will be conducted in two parts: a phase I study and a phase II study. In both instances, a treatment cycle is 28 days (4 weeks). Subjects will take OSI-906 by mouth, twice a day, every day. Subjects will receive gemcitabine through an IV in clinic over 30 minutes on days 1, 8 and 15 of each 28-day cycle. Subjects will take erlotinib by mouth, once a day, every day.

At every visit subjects will have a physical exam and blood tests. An EKG will be done on days 1, 8 and 15 of cycle 1 and on day 1 of all subsequent cycles. A CT scan will be done every 2 cycles (8 weeks).

Subjects will complete a daily drug diary and perform glucose monitoring (finger stick) once daily at home.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic ductal adenocarcinoma
* Measurable disease
* Life expectancy > 12 weeks
* Normal organ and marrow function
* Fasting blood glucose </= 150 mg/dL
* Able to swallow pills

Exclusion Criteria:

* Prior chemotherapy or radiotherapy for treatment of pancreatic cancer
* Receiving any other experimental agent
* Known brain metastases
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to gemcitabine, erlotinib, or OSI-906
* Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, or diarrhea)
* Use of enzyme-inducing anti-epileptic drugs
* Diabetes mellitus which requires the use of exogenous insulin for glucose control
* Major surgery within 4 weeks of the start of study treatment
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Use of strong or moderate CYP1A2 inhibitors/inducers
* Pregnant or breast feeding
* History of a different malignancy unless disease-free for at least 3 years
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 1 years
  Phase I study to assess the safety, tolerability and maximally tolerated dose (MTD) of OSI-906 administered in combination with gemcitabine and erlotinib is patients with metastatic pancreatic ductal adenocarcinoma
Survival among patients receiving gemcitabine + erlotinib versus gemcitabine + erlotinib + OSI-906 | 2 years
  Phase II trial to assess overall survival associated with OSI-906, gemcitabine and erlotinib compared with gemcitabine and erlotinib alone in patients with previous untreated metastatic pancreatic ductal adenocarcinoma

SECONDARY OUTCOMES:
Progression-free survival among patients receiving gemcitabine + erlotinib vs. gemcitabine + erlotinib + OSI-906 | 2 years
  To assess progression-free survival associated with OSI-906, gemcitabine and erlotinib compared to gemcitabine and erlotinib alone in patients with previously untreated metastatic pancreatic ductal adenocarcinoma
Tumor response rate among patients receiving gemcitabine + erlotinib versus gemcitabine + erlotinib + OSI-906 | 2 years
  To assess tumor response rate associated with OSI-906, gemcitabine and erlotinib compared to gemcitabine and erlotinib alone in patients with previously untreated metastatic pancreatic ductal adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Brian Wolpin, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts